CLINICAL TRIAL: NCT06665282
Title: Efficacy of Pulsed High Intensity Laser Therapy in Treatment of Psoriatic Hand Arthritis
Brief Title: Efficacy of Pulsed High Intensity Laser Therapy in Psoriatic Hand Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Shawky Helmy Abdelhamid, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mahmoud-004436
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: High Intensity Laser Therapy; Psoriasis; Hand
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed high intensity level laser therapy group (Experimental): This group includes 38 patients who will receive pulsed high intensity level laser therapy 3 sessions per week over 8 successive weeks in addition to routine physical therapy in the form of hot therapy, stretching and strengthening exercises
  Interventions: Device: Pulsed high intensity laser therapy; Other: Routine physical therapy program
- Shame pulsed high intensity laser level therapy (Active Comparator): This group includes 38 patients who will receive shame pulsed high intensity laser level therapy 3 sessions per week over 8 successive weeks in addition to routine physical therapy in the form of hot therapy, stretching and strengthening exercises
  Interventions: Device: sham pulsed high intensity laser therapy; Other: Routine physical therapy program

INTERVENTIONS:
Device: Pulsed high intensity laser therapy — The study employs a BTL-6000 high-intensity laser therapy (12 W) to apply high intensity laser therapy to deep tissues. high intensity laser therapy therapy uses powerful beams (>500 mw) to penetrate deeper, delivering high multi-directional energy in a short time. Pulsed laser therapy, a form of high intensity laser therapy therapy, enhances cell metabolism without disrupting it.
  High-intensity laser therapy is a safe treatment method consisting of three phases. The first phase involves fast scanning around the wrist, hand, and fingers, with fluencies set at 510, 610, and 710mJ/cm2. The second phase involves holding the handpiece vertically to 90° on 10 fixed points around the metacarpophalangeal and interphalangeal joints, each radiated for 15 seconds, and a total dose of 1500 J. The third phase is the same but at a slower rate, with a total energy of 300 J.
  Arms: Pulsed high intensity level laser therapy group
Device: sham pulsed high intensity laser therapy — Patients in the control group will receive sham high-intensity laser therapy, where all parameters will be set up without switching on the start button and high intensity laser therapy machine is switched on with a visible light beam only
  Arms: Shame pulsed high intensity laser level therapy
Other: Routine physical therapy program — All patients of the study and control groups will receive the same routine physical therapy program for 30minutes and three times per week for successive eight weeks in the form of hot therapy, stretching and strengthening exercises. Hot therapy, in the form of warm baths for 10minutes, is applied before stretching exercises on the wrist joint and fingers to relieve joint pain and increase the range of motion. Strengthening exercises are in the form of isometric exercise for hand muscles and fingers to maintain muscles strength and joints flexibility

SUMMARY:
The purpose of the study was to evaluate the therapeutic efficacy of pulsed high intensity level laser therapy in improving symptoms of psoriatic hand arthritis.

DETAILED DESCRIPTION:
Psoriatic arthritis is a chronic, inflammatory joint disease affecting 20%-30% of patients with psoriasis. It affects peripheral joints and axial skeleton, causing pain, stiffness, swelling, and joint destruction. High-intensity laser therapy can control inflammation and improve pain relief, range of motion, and functional improvement. This study aims to examine High-intensity laser therapy efficacy in managing Psoriatic arthritis, aiming to provide a safe, effective, and noninvasive treatment method.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes of patients their age range between 30-50 years.
* Bilateral PsA following psoriasis
* All participants who are diagnosed with PsA, and experience clinical symptoms such as pain, swelling, tenderness and stiffness less than 1 year from the beginning of disease.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* Positive rheumatic factor
* Circulatory disorders
* Diabetes
* Pregnant woman
* Skin diseases like urticaria.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of change of Hand Grip Strength using manual dynamometer | at baseline and after 2 months
  The Handheld Jamar dynamometer device 12-0600 will be used to measure hand grip strength, with a readout in pounds and kilograms. The strength will be measured with the elbow at 90° according to the American Society of Hand Therapists' recommendations. Patients will be instructed to sit while the affected limb is placed in shoulder adduction, internal rotation, elbow flexion, forearm mid position, and wrist neutral position. Three consecutive measurements will be performed with a 2-minute interval, and the mean strength value of the three trials will be considered as the hand grip measure.

SECONDARY OUTCOMES:
assessment of Joint counts for tenderness | at baseline and after 2 months
  Joint counts for tenderness was the sum of the number of the affected joints
assessment of Joint swelling count | at baseline and after 2 months
  Joint swelling count is the sum of the swollen joints at the dominant hand before and after the treatment
assessment of pain intensity using visual analogue scale | at baseline and after 2 months
  The Visual Analog Scale was used to measure pain intensity, with a 100mm horizontal line starting with no pain and ending with worse pain. Patients marked their pain intensity points on the scale, and the researcher measured the distance between the "no pain" mark and the patient's mark, providing a range of scores from 0 to 100mm.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt